CLINICAL TRIAL: NCT06246474
Title: Impact of Kinesio Taping on Kyphosis and Quality of Life in Adolescents
Acronym: kinesio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa abd elmohsen ali, PHD student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004905; P.T.REC/012/004905 (Other: Cairo University)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Kyphosis; Kyphosis Thoracic; Kyphosis Postural Thoracic
Keywords: kyphosis; postural kyphosis; Forward head posture; Adolseccent
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (A) (No Intervention): Adolescents in control group (A) will received a designed physical therapy program for the treatment of thoracic kyphosis
- group (B) (Experimental): Adolescents in study group (B) will received the same designed physical therapy program for the control group in addition to Kinesio taping.
  Interventions: Procedure: physical therapy program

INTERVENTIONS:
Procedure: physical therapy program — Arm Description: Adolescents in study group (B) will received the same designed physical therapy program for the control group in addition to Kinesio taping.
  Other Names: Kinesio taping
  Arms: group (B)

SUMMARY:
Kyphosis, a posture disorder, is excessive curvature of the thoracic area in the spine. In a healthy person, there is a normal kyphosis angulation in the thoracic and sacral areas in the sagittal plane. Since the sacral area is more stable, pathological conditions generally occur in the thoracic area.

Kyphosis causes a bowing of the back, which leads to a hunchback or slouching posture. Normal values for the thoracic kyphosis are between 20˚ and 40˚ of angulations. When the curve of the thoracic spine exceeds this, it is described as either a postural kyphosis or Scheuermann's kyphosis.

The study question is: Does kinesio taping have an effect on kyphosis and quality of life in adolescents?

DETAILED DESCRIPTION:
The purpose of the study is to determine the effects of kinesio taping on:

* Kyphotic curve.
* Forward head posture.
* Quality of life in adolescents. Postural kyphosis is the most common type that causes slouching in thoracic curve can occur in young age, it can be called 'slouching' and is reversible by correcting muscular imbalances.

Adolescent's kyphosis curve appear by bad habitual postures due to a carry-over effect from temporary changes in posture during computer use and smart phones.

Forward head posture (FHP) is characterized that cervical spine is held in protracted position for prolonged duration, it can lead to alterations in head posture ultimately leading to poor posture which is thought to be a deviation from neutral or normal posture.

Failure of the head to align with the vertical axis of the body can lead to further malalignments in the body, namely, rounded shoulders and increased thoracic kyphosis, to compensate for the altered location of the LOG, leading to further impairments . A combination of all these postural deviations is often known as "slouched posture" or "slumped posture." The Kinesio taping method was applied to correct the alignment of weak muscles as well as facilitating joint motion as a result of the tape's recoiling qualities. It was designed to be the approximate thickness and elasticity of skin and be worn three to five days at a time.

Kinesio taping is a therapeutic tool used with increasing frequency within musculoskeletal rehabilitation and to maintain preferred body alignment. It is a complementary treatment and is designed to facilitate the body's natural healing, Process while allowing support and stability to 5 muscles and joints without restricting the body's range of motion.

Due to the lack of research area of kinesio taping on kyphosis in adolescents, So, the purpose of the study is to know impact of the Kinesio taping on kyphosis and quality of life in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Their age will be ranged from 15 to 18 years.
* They will have forward head posture.
* They will have postural kyphosis with Cobb's angle more than 45 degree.
* Their body mass index of female adolescents will be ranged between (19.5 - 20.7)

Exclusion Criteria:

* Visual or hearing defects.
* Congenital anomalies in spine region.
* Fractures of upper limb.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
cobbs angle x-ray for selection of the patient | 2 months
  Full length AP (anterior/ posterior, front/ back ) film x-ray will be taken of the spinal column ,these x- rays will be used to determine curve flexibility and evaluate vertebral wedging and end plate irregularities
inclinometer for selection patients of kyphotic curve measurements | 2 months
  Two gravity-dependent inclinometers (Isomed, Inc, USA) will be used. The feet of the inclinometers were 2.5 cm apart, which remained constant for all subjects, manual inclinometer probes, the two MEMS sensors are mounted 90 degree
modified baseline goniometer for FHP angle's measurement | 2 months
  The modified goniometer is a simple and cost-effective modification of the universal goniometer; it has an excellent reliability and validity method for objectively assessing forward head posture.
quality of life questionnaire (PEDS) for quality of life | 2 months
  Pediatric Quality of Life Inventory (PedsQL) Module3.0 will be used to assess QOL of all adolescents. Arabic version will be used in this study (Shemy et al., 2019) (Appendix III). The parent will be asked about the grade of the problem of each item that the adolescents had in the past month.
Tape measurment for chest expansion range of motion. | 2 months
  Tape measurment for chest expansion range of motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Due to University rules